CLINICAL TRIAL: NCT00736827
Title: BK Virus and Renal Dysfunction in Postoperative/Posttraumatic Critically Ill Patients
Acronym: BICUK
Status: Completed | Type: Observational
Sponsor: University of Ulm (Other)
Collaborators: University of Wuerzburg (Other)
Responsible Party: Principal Investigator, Manfred Weiss, Professor, MD, MBA, University of Ulm
Other Study IDs: Anae_ICU_Ulm_BKV
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Acute Renal Failure; SIRS; Sepsis; Critically Ill; Multiple Organ Dysfunction Syndrome
Keywords: BK virus; acute renal failure; hemodiafiltration; humans; patients; polytrauma; surgery; complement; inflammation; inflammatory response; biomarkers; cytokines; cell surface markers; functional polymorphisms; infections; systemic inflammatory response syndrome; SIRS; sepsis; severe sepsis; shock; organ dysfunctions; SOFA; severity of disease; APACHEII; SAPSII; SPAPS3; length of stay; outcome; mortality
MeSH Terms: conditions — Acute Kidney Injury; Sepsis; Critical Illness; Multiple Organ Failure; Multiple Trauma; Inflammation; Infections; Systemic Inflammatory Response Syndrome; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, white blood cells; urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with non-septic shock: Postoperative/posttraumatic surgical critically ill patients with non-septic shock with threatening acute renal failure
- Patients with septic shock: Postoperative/posttraumatic surgical critically ill patients with septic shock with threatening acute renal failure

SUMMARY:
The purpose of this study is to find out whether acute renal failure is associated with BK virus reactivation in postoperative/posttraumatic critically ill patients with severe SIRS/sepsis and shock.

DETAILED DESCRIPTION:
Polyomavirus BK virus (BKV) infection and nephropathy is a significant cause of allograft dysfunction in kidney transplantation. Clinical manifestation ranges from BK viremia and nephritis to renal dysfunction. It has been suggested that BK virus reactivation alone is not sufficient to cause BK viremia and nephropathy, thus a second hit is essential for kidney specific damage, such as an inflammatory reaction or ischemia. Critically ill postoperative/posttraumatic patients via the systemic inflammatory response syndrome (SIRS) and the compensatory antiinflammatory response syndrome (CARS) are at increased risk to develop organ dysfunctions, such as acute renal failure. CARS, reflecting postoperative/posttraumatic immunosuppression, may favor viral reactivation. However, prevalence of BK viremia in critically ill postoperative/posttraumatic patients has up to now not been systematically evaluated. Moreover, it is not known whether BK viremia is associated with a distinct biomarker pattern in these patients. Therefore, the present study is performed to clarify whether postoperative/posttraumatic immunosuppression is associated with BK viremia, and acute renal failure with BK virus reactivation, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill, postoperative/posttraumatic patients with threatening acute renal failure

Exclusion Criteria:

* Life expectancy < 24 hours
* Participation in other trials
* Known or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative/posttraumatic critically ill patients admitted to the intensive care unit
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2008-08; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Association between BK virus reactivation and acute renal dysfunction | Daily monitoring of acute renal failure, first day of acute renal dysfunction, first days on hemodiafiltration, first day after hemodiafiltration, before demission from intensive care unit or death.

SECONDARY OUTCOMES:
Pattern of biomarkers and surface markers on leukocytes. | First day of acute renal dysfunction, first days on hemodiafiltration, first day after hemodiafiltration, before demission from intensive care unit or death.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Weiss, MD, MBA, Principal Investigator — University Hospital Ulm
Locations (1):
- Clinic of Anesthesiology, Ulm, Germany

REFERENCES:
- [Result] Nass M, Weissbrich B, Huber M, Schneider EM, Weiss M. BK viremia in critically ill surgical patients with hemorrhagic or septic shock. BMC Res Notes. 2012 Feb 16;5:100. doi: 10.1186/1756-0500-5-100. PMID 22339896
- See also: Nass M, Weissbrich B, Huber M, Schneider EM, Weiss M. BK viremia in critically ill surgical patients with hemorrhagic or septic shock. BMC Research Notes 2012; 5:100 (16 Februar 2012). doi:10.1186/1756-0500-5-100 — http://www.biomedcentral.com/1756-0500/5/100